CLINICAL TRIAL: NCT06779045
Title: A Phase 1,Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of AK-1286 in Patients With Advanced Solid Tumors
Brief Title: A Study of AK-1286 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK-1286-001
Record Dates: First submitted 2025-01-02; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK-1286 (Experimental): After a screening period of approximately 28 days, eligible patients will receive oral YL-15293 once or twice daily until documented disease progression, unacceptable AEs, intercurrent illness prevents further administrations of study treatment, investigator's decision to withdraw the patient, the patient withdraws consent, pregnancy of the patient, or for administrative reasons. Following the end of treatment, patients will continue to be followed for safety for 30 days. Patients who permanently discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.
  Interventions: Drug: AK-1286

INTERVENTIONS:
Drug: AK-1286 — Cohort 1: 1 mg/d QD AK-1286 PO,DLT observation period: 21 days. Cohort 2: 2 mg/d BID AK-1286 PO,DLT observation period: 21 days. Cohort 3: 4 mg/d BID AK-1286 PO,DLT observation period: 21 days. Cohort 4: 5 mg/d BID AK-1286 PO,DLT observation period: 21 days. Cohort 5: 16 mg/d BID AK-1286 PO,DLT observation period: 21 days. Cohort 6: 24 mg/d BID AK-1286 PO,DLT observation period: 21 days. Cohort 7: 36 mg/d BID AK-1286 PO,DLT observation period: 21 days. Cohort 8: 50 mg/d BID AK-1286 PO,DLT observation period: 21 days.

SUMMARY:
This is a phase 1 open label multicenter study to evaluate the maximum tolerance, safety, tolerance and PK of AK-1286 in patients with advanced solid tumors, so as to confirm the recommended phase 2 dose of AK-1286 and obtain the preliminary efficacy information of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years (including cut-off value), gender is not limited;
* Patients with histologically or cytologically diagnosed advanced malignant solid tumors who have failed or are unable to tolerate standard treatment regimens with systemic standard therapy.
* participants in the dose expansion phase must have quantifiable lesions according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
* Anticipated minimum survival duration of 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must meet the laboratory criteria.A. Bone marrow function needs to meet#ANC≥1.5×109/L#PLT≥100×109/L#Hb≥9g/dL B. renal function#Cr≤1.5 times the upper limit of normal value#or Creatinine clearance≥50ml/min C. liver function#total bilirubin<1.5 x ULN#For subjects with documented Gilbert syndrome,< 2.0 x ULN or subjects with indirect bilirubin levels suggesting a source of extrahepatic elevation<3.0 x ULN#ALT and AST≤ 2.5 x ULN#If liver metastasis occurs≤ 5 x ULN#D. Coagulation function#Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper normal limit (ULN), or international normalized ratio (INR) < 1.5 or within the target range (if preventive anticoagulant therapy is performed# E). The corrected QT interval (QTcF) of Fridericia method is less than 450 ms for males and less than 470 ms for females.
* The elution period of macromolecular drugs is ≥ 4 weeks, and that of oral fluorouracil and small molecule targeted drugs is ≥ 2 weeks
* Fertile women must have a negative blood pregnancy test within 7 days before receiving the first study drug;
* For fertile men and women, they must be willing to use appropriate contraceptive methods 30 days before the first study drug administration and 120 days after the last study drug administration;
* Did not participate in the clinical trial as a subject within 1 month before participating in the trial;
* According to the judgment of the researcher, the compliance is high,willing to complete the test and can abide by the test scheme;
* Voluntarily participate in this clinical trial, understand the research procedures and be able to sign the informed consent form in writing.

Exclusion Criteria:

* Untreated patients with brain metastasis
* Other malignant tumors in recent five years. Basal cell carcinoma of the skin, except squamous cell carcinoma of the skin or cervical carcinoma in situ after potential treatment;
* Myocardial infarction, symptomatic congestive heart failure (New York Heart Association > grade II), unstable angina pectoris or arrhythmia requiring drug treatment occurred within 6 months before enrollment;
* Have a history of gastrointestinal diseases or gastric surgery or inability to swallow oral drugs;
* Active infection requiring treatment;
* Patients with active hepatitis B (hepatitis B surface antigen and / or hepatitis B core antibody positive and HBV-DNA > 103 copies /mL or 200IU/mL) or hepatitis C patients (hepatitis C virus positive and / or HCV-RNA positive) or HIV positive patients are required to receive treatment.
* Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks before the first use of the study drug, or elective surgery during the trial, or therapeutic or palliative radiotherapy within 2 weeks before the first use of the study drug;
* Allergic constitution, or known history of allergy to this drug component;
* According to the researchers' judgement, there are serious diseases that may endanger the safety of patients or affect the completion of research, such as uncontrollable hypertension, uncontrollable diabetes and thyroid diseases.
* There is fluid accumulation in the third space that cannot be controlled by drainage or other methods (such as massive identification and hydrothorax)
* Have a clear history of neurological or mental disorders；
* The researchers believe that the subjects are not suitable to participate in this study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of drug limited toxicities (DLTs) | From Time of First dose through DLT observation period, 21 days
  To assess by the occurrence of Drug Limited Toxicities (DLTs)
Incidence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  To assess by the occurrence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs)
Number of patients with changes in laboratory parameters from baseline | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  To assess safety of AK-1286
Number of participants with changes in clinically significant vital sign from baseline | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  To assess safety of AK-1286

SECONDARY OUTCOMES:
The overall response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The overall response rate (ORR) will be estimated based on the proportion of evaluable patients whose overall response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1.response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1
Progression free survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS, defined as the time from the first dose of study treatment to The tumor progresses for the first time
Overall survival（OS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The time from randomization to death for any reason
Disease control rate（DCR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The percentage of cases with remission (PR+CR) and stable lesions (SD) after treatment

IPD SHARING:
Plan to Share IPD: No